CLINICAL TRIAL: NCT06758011
Title: Feasibility Study for ivWatch® in Prevention of Extravasation of Vesicants in an Oncology Setting
Brief Title: ivWatch in Prevention of Extravasation of Vesicants in an Oncology Setting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I-2794222
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Oncology; Extravasation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Medical Device Usage (Experimental): Patients utilize ivWatch device at time of already scheduled chemotherapy on study
  Interventions: Device: ivWatch

INTERVENTIONS:
Device: ivWatch — Patients wear ivWatch device at time of already scheduled chemotherapy on study.

SUMMARY:
This study aims to determine the feasibility of using the ivWatch (registered trademark) device to determine if there is an infiltration at the site of a peripheral intravenous (PIV) catheter. An infiltration is when the IV fluid leaks out of a vein and into the surrounding tissue. If medication starts leaking outside the vein, it can cause damage to the surrounding tissue. Using the ivWatch device may identify leaking fluid before the nurse is able to visually observe the signs or symptoms of the leaking fluid.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of using the ivWatch device to detect extravasations of peripheral vesicants given in an adult oncology ambulatory population.

SECONDARY OBJECTIVE:

I. Evaluate the clinical outcomes of extravasations that occur with the use of the ivWatch device.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a peripheral IV for infusion of vesicant or vesicant-like agents (chemotherapy, other vesicant medications).
* PIV must be inserted
* Participant (or legal representative) must understand the nature of this study and verbally consent with the Research Study Information Sheet prior to receiving any study related procedure

Exclusion Criteria:

* Patients who are not getting a vesicant, irritant or vesicant like fluid infused.
* Patients who are bruised, scarred, or tattooed in the area of the PIV.
* Patients with skin integrity issues at the site of the PIV.
* Patients who are on "light precautions."
* Not for use in power injectors.
* Not for use on mediports, implanted ports, IVAD, central lines, PICC lines.
* Patients without a cancer diagnosis.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-11-17 (Estimated)

PRIMARY OUTCOMES:
Ratio of number of ivWatch devices used for vesicant therapy | Up to 1 year
  the ratio of number of the device used for vesicant therapy over the total number of vesicant therapies for study participants

SECONDARY OUTCOMES:
Change in number of extravasations while wearing ivWatch | Up to 1 year
  Summary of patient level data will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States